CLINICAL TRIAL: NCT04512222
Title: EARLY-MYO-AF (EARLY Integrated Therapies on MYOcardial Function Improvements in Patients With Atrial Fibrillation) Registry
Brief Title: EARLY-MYO-AF Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY-MYO-AF
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2012-01

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry is to depict the myocardial function improvement in AF patients by integrated therapy and to assess the prognostic discrepancies of various intervention modalities. Information will be collected prospectively in about 5000 AF patients. Subjects will be followed for up to 3 years.

DETAILED DESCRIPTION:
This is a prospective, single-centered, non-randomized, observational registry study of AF patients that undergo radio-frequency catheter ablation, left atrial appendage occlusion or surgical ablation. Information of other medication intervention and clinical outcomes are also prospectively collected in the database. This project will establish a prospective registry of 5000 AF patients with follow-ups of up to 3 years.

The aim of the project will be as following:

1. To investigate pathophysiological changes of both atrial and ventricular myocardial function in AF patients.
2. To identify clinical indices (including baseline, comorbidities, medication or operational interventions) that are associated with adverse clinical outcomes.
3. To spot potential therapeutical targets in the continuum of AF: from risk-factors elimination to mortality and disability prevalence reduciton.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must be at least 18 years old at the time of enrollment.
* Patients who are clinically indicated catheter ablation or other interventions (LAAC or surgical maze procedure) for persistent or long standing persistent AF.

Exclusion Criteria:

* Contraindication for anticoagulation therapy
* Another (non-AF) indication for long term anticoagulation
* Patients who have been enrolled as a respondent on other clinical studies
* Inability to attend scheduled, periodic office visits for follow-up
* Pregnancy
* Patient has a life expectancy of less than 6 months due to any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients undergo interventional or surgical procedures are eligible for this registry.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 3 years
  A composite of stroke/transient ischemic attack, thromboembolism and all-cause mortality.

SECONDARY OUTCOMES:
Major bleeding | 3 years
  A composite of events listed below: a)Bleeding resulting in a decrease in hemoglobin of ≥2 g/dL or over a 24-hour period b) Bleeding leading to a transfusion of 2 or more units of packed red blood cells c) Bleeding that occurs in a critical site (intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome or retroperitoneal) d. Bleeding that leads to death.

OTHER OUTCOMES:
Atrial fibrillation event | 3 years
  Documented Atrial fibrillation of more the 5 minutes duration.

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Wang, Prof., Study Chair — Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang XH, Kong LC, Shuang T, Li Z, Pu J. Macro-reentrant atrial tachycardia after tricuspid or mitral valve surgery: is there difference in electrophysiological characteristics and effectiveness of catheter ablation? BMC Cardiovasc Disord. 2021 Nov 12;21(1):538. doi: 10.1186/s12872-021-02368-w. PMID 34772362